CLINICAL TRIAL: NCT06957769
Title: Biological Impacts of Rising Temperatures on Maternal, Fetal, and Newborn Health: A Cohort Study (BIRTH Cohort)
Acronym: BIRTH
Status: Recruiting | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dr Jai Kumar Das, Doctor, Aga Khan University
Other Study IDs: 2025-8888-34528; 227190/Z/23/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2025-05-02; First posted 2025-05-04 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Low Birth Weight Baby; Small for Gestational Age (SGA); Preterm Birth; Pregnancy Complications; Birth Outcome, Adverse; Heat Strain; Infant Morbidity; Infant Mortality; Neonatal Mortality
Keywords: heat stress; high ambient temperature; climate change; birth outcomes; pregnancy; cohort study; Pakistan
MeSH Terms: conditions — Premature Birth; Pregnancy Complications; Infant Death; Heat Stress Disorders | interventions — Heat-Shock Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For the sub-cohort of 1000 women, nasopharyngeal swabs and stool samples will be retained during pregnancy. At delivery. their placental samples will be retained. Breastmilk sampling will be done in first six months after delivery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnancy cohort: Pregnant women, more than 18 years of age and residents of study sites Matiari, Tharparkar and Tando Muhammad Khan
  Interventions: Other: heat stress

INTERVENTIONS:
Other: heat stress — Heat stress (exposure) will be quantified using validated environmental heat stress indices, including the mean Heat Index (HI). The heat index represents the apparent temperature or how hot it feels to the human body when air temperature is combined with relative humidity. Individual-level ambient temperature heat exposure will be assessed using wearable temperature and humidity loggers.

SUMMARY:
The goal of this study is to learn how being exposed to high environmental temperatures during pregnancy affects the health of pregnant women and their babies. The study also aims to understand how the body responds to heat stress during pregnancy and how this might lead to pregnancy complications and birth problems like early birth or low birth weight.

The main questions that the study aims to answer are:

1. What are the acute and chronic effects of environmental heat exposure on pregnancy and birth outcomes across different trimesters?
2. Through which biological pathways does heat stress impact maternal, fetal, and infant health across varying gestational ages?
3. How do socio-demographic factors, maternal characteristics, and nutritional status of women modify the relationship between environmental heat exposure and adverse pregnancy outcomes?

The study will take place in rural parts of Sindh, Pakistan. These areas often experience extreme heat and have limited access to electricity or cooling systems like fans or air conditioners.

This study will include pregnant women who are in their first trimester (under 14 weeks of pregnancy). Before starting any study activities, researchers will explain the study to each woman in a language she understands and ask for her written permission to take part (informed consent).

At the beginning of the study, participants will visit a study clinic. During this visit, researchers will check their height and weight, perform an ultrasound, and collect a small amount of blood for testing. Participants will also be asked to wear a small device that measures the air temperature and humidity in their surroundings.

The researchers will follow each participant during her pregnancy, with visits during the second and third trimesters at the study clinic. At each visit, researchers will check how much heat the participant has been exposed to using the data from the device and from her own answers to a simple questionnaire. The questionnaire will have questions about their heat exposure at work, home, type of clothing, and how they deal with hot weather. Serial ultrasound, blood and urine tests will be conducted so researchers can study signs of stress, hydration, and other changes in the body. A smaller group of participants will also wear a device to measure their body skin temperature, heart rate, physical activity and sleep during pregnancy.

When the baby is born, researchers will collect information about the birth, including the baby's weight and length, the time of delivery, and whether there were any complications during birth. After delivery, both the mother and baby will be followed for up to 12 months. During this time, the research team will check the health of both the mother and baby and see how heat exposure during pregnancy may affect the baby's growth over time. At delivery, placental weight and volume will be collected for a smaller group of women. Breastmilk sampling will also be done for this group of women to understand the effect of high temperatures on breastmilk quality.

This study does not involve any treatment or medicine. Instead, researchers will observe the participants to learn how real-life heat exposure affects them during pregnancy. The findings from this study may help public health officials and governments find better ways to protect pregnant women and babies from the harmful effects of climate change and extreme heat, especially in places with limited resources.

DETAILED DESCRIPTION:
Background

Anthropogenic climate change has led to a significant rise in global temperatures, resulting in more frequent, intense, and prolonged heat events. This has profound health implications for vulnerable populations, particularly in low-resource settings. Pregnant women are particularly susceptible, as heat exposure can disrupt maternal thermoregulation and fetal development, potentially leading to complications such as preeclampsia, gestational diabetes, hypertensive disorders, cardiovascular events, and increased risks of preterm birth, low birth weight (LBW), small-for-gestational-age (SGA) births, and stillbirths.

Studies have indicated a 1.04-fold increase in preterm birth odds per 1°C rise in temperature, with even greater risks during heatwaves. Additionally, associations have been observed between heat exposure and stillbirth, congenital anomalies, and gestational diabetes. Despite growing epidemiological evidence, there is limited data on the biological mechanisms driving these associations, particularly in low- and middle-income countries (LMICs).

Several biological pathways have been proposed to explain the impact of heat on pregnancy and birth outcomes. These include heat-induced hyperthermia in early pregnancy associated with neural tube defects. Exposure to high temperatures may lead to placental insufficiency due to altered blood flow. Chronic uteroplacental insufficiency may cause fetal hypoxia and intrauterine growth retardation (IUGR) and small for gestational age (SGA) newborns. Other heat stress-related pathways include oxidative stress, inflammatory responses, and prostaglandin-mediated change. In late pregnancy, heat exposure may induce early labor and preterm birth through release of oxytocin and prostaglandins. Increased maternal core temperature can impair fetal oxygenation and growth by redistributing blood flow away from the uterus.

Study Rationale

Despite growing concern over the impact of extreme heat on maternal and fetal health, evidence on the biological pathways in humans remains sparse and inconsistent, largely due to challenges in isolating heat stress as an independent exposure during pregnancy. While animal studies and limited human experimental research have identified physiological changes under heat stress, the specific pathophysiological mechanisms linking heat exposure to adverse pregnancy and birth outcomes in humans remain poorly understood. Notably, most available evidence stems from high-income countries, despite the fact that the burden of preterm birth, stillbirth, and fetal growth restriction is disproportionately higher in low- and middle-income countries (LMICs).

This study aims to address these gaps by exploring the potential biological pathways linking heat exposure to adverse maternal and birth outcomes in a high-risk LMIC setting. In the Sindh province of Pakistan, where this study is based, pregnant women are frequently exposed to extreme temperatures both outdoors and indoors. They often engage in manual agricultural work, care for livestock, and perform household chores like cooking over open fires, often without access to cooling mechanisms. These intersecting vulnerabilities-physical exertion, prolonged heat exposure, and limited structural protection-contribute to their heightened risk.

Study Objectives

The primary objectives of the study are:

* To assess the acute and sustained effects of environmental heat exposure on pregnancy and birth outcomes in rural and peri-urban areas of Pakistan.
* To assess the bio-physiological pathways through which heat stress affects maternal, fetal, and infant health across different gestational ages in rural and peri-urban areas of Pakistan.

The secondary objectives are:

• To evaluate how gestational age, socio-demographic, maternal and nutritional factors modify the association between heat exposure and adverse pregnancy outcomes in rural and peri-urban areas of Pakistan.

METHODS

Study Design and Study Sites

A prospective cohort study will be conducted among pregnant women residing in three districts of Sindh province of Pakistan: Matiari, Tando Muhammad Khan (TMK), and Tharparkar. These regions experience extreme summer temperatures and face multiple socio-economic challenges, including poor infrastructure, food insecurity, and high rates of maternal and neonatal health complications. Participants will be enrolled in their first trimester and followed through delivery and up to 12 months postpartum. The study will integrate environmental measurements, wearable sensors, imaging studies and biological samples to assess physiological, behavioral, and environmental responses to heat stress.

Sample Size

To detect a 15% increase in the risk of LBW among pregnant women exposed to heat stress compared to an unexposed cohort (1:2 ratio), and assuming 80% power, a 5% significance level, and a 20% attrition rate, 6,000 participants will be required. This calculation is based on a baseline LBW prevalence of 26.2% reported in the 2018 National Nutrition Survey for the rural population. The sample size for SVN under the same assumptions is 2,106 based on a prevalence of 46%.

For the detailed sub-study, sample size calculations were based on various key physiological parameters assessed in controlled settings, including changes in skin temperature, maternal heart rate, blood pressure, cardiac output, and fetal heart rate. To detect a 10% change in these parameters, the maximum required sample size is 200 participants, assuming 90% power, a 5% significance level, and a 20% attrition rate. However, due to the limited scope of previous studies conducted under controlled conditions and the anticipated higher attrition rate, we have chosen a sub-study sample size of 1,000 women.

Participant Recruitment and Enrollment

Pregnant women will be identified through community-based outreach in coordination with Lady Health Workers (LHWs). Field teams will conduct site mapping and community engagement to identify women who are newly married, within 1-2 years of their last pregnancy, or planning conception. Pregnancy status will be confirmed through rapid urine tests, followed by ultrasound verification conducted by study physicians at designated study offices.

After obtaining informed consent, a recruitment form will be completed. At study offices, antenatal assessment, ultrasound imaging, and biological sample collection will be performed. For the sub-study on physiological monitoring, a subset of participants will be enrolled based on their consent to wear wearable devices and allow skin temperature assessment. Transportation assistance will be provided to facilitate participation in study activities.

Data Collection Procedures

Baseline Assessments

At enrollment, gestational age will be estimated using fetal crown-rump length via ultrasound, based on the INTERGROWTH-21st protocol (±7 days accuracy). Baseline data will include sociodemographic information, medical and obstetric history, housing characteristics, occupational exposure, and anthropometric measurements. A standardized 24-hour dietary recall will be conducted at each antenatal care (ANC) visit, capturing information on food intake, frequency, meal composition, and seasonal variations.

Follow-Up Assessments

Serial ultrasounds will be conducted at 12-14, 18-22, 28-32, and 36-37 weeks' gestation, including Doppler and fetal echocardiography. Maternal blood and urine samples will be collected to assess markers such as complete blood count (CBC), hemoglobin, ferritin, glucose tolerance, dehydration status, and biological stress indicators. Samples will be handled using standardized protocols, transported in temperature-controlled containers (2-8°C), and stored at the Aga Khan University Nutrition Research Laboratory (NRL), Karachi, for analysis.

Environmental Exposure Monitoring

Ambient indoor temperature will be recorded continuously using wearable temperature/humidity loggers. Wet Bulb Globe Thermometers will provide outdoor environmental indices, accounting for multiple heat stress factors (e.g., radiant temperature, humidity, wind speed, radiation and clothing) and to calculate WBGT for each participant throughout their pregnancy.

A subset of participants will wear smartwatches to monitor heart rate, sleep patterns, and physical activity throughout pregnancy. Skin temperature will be recorded using i-Button loggers worn in customized abdominal belts. A field team will oversee device function and data transfer fortnightly.

Delivery and Postnatal Follow-Up:

At delivery, newborn weight, length, mid-upper arm circumference (MUAC), and head circumference will be recorded by trained staff within 48 hours of birth. A delivery notification system and routine calls when the participant is near term will ensure timely outcome capture.

For the sub-cohort, placental tissue and cord blood will be collected within 10-15 minutes post-delivery, snap-frozen, and stored at -80°C. Additional bio-specimens (stool and sputum) will be archived for future analyses, including epigenetic and molecular analyses. Breastmilk sampling will also be done for the sub-cohort to understand the effect of high temperatures on breastmilk quality and composition.

The mother-infant dyad will be followed for twelve months post-delivery, with monthly assessments of anthropometry, feeding practices, immunization, morbidity, and neurodevelopment.

Key maternal and newborn health outcomes will be tracked, including pregnancy complications, gestational age at delivery, birth weight, infant growth, and maternal and neonatal mortality.

Training of Study Staff and Quality Assurance

Experienced local personnel, including physicians, sonologists, nurses/ midwives, and data collectors, will be hired. Study doctors will have prior obstetrics and gynecology training, and experience in obstetric ultrasound. They will receive a 3-month training in ultrasound and maternal echocardiography at Aga Khan University (AKU), alongside completion of the International Society of Ultrasound in Obstetrics and Gynecology (ISUOG) ultrasound course.

Each study site will have three teams (two data collectors and one supervisor per team). Centralized training will include orientation to the study protocols, a question-by-question tool review, and anthropometry training per Food and Nutrition Technical Assistance III (FANTA III) guidelines. Field practice and pilot study will be conducted. Personnel operating the wearable devices will receive additional training in handling the devices and regular data retrieval.

Maternal and infant anthropometry will follow INTERGROWTH-21st standards. Maternal weight will be measured with Seca 874 U scales (precision: 0.1 kg). Newborn weight will be recorded within 48 hours using Seca 354 infant scales. Infant recumbent length will be measured with an Infantometer; head circumference and MUAC will be recorded to the nearest millimeter. All equipment will be calibrated biweekly. Maternal weight will be recorded twice by the same anthropometrist, and infant measurements will be taken independently by two blinded anthropometrists.

Statistical Analysis

Ambient heat exposure during pregnancy for each participant will be assessed using Mean Heat Index calculated from wearable temperature and humidity loggers using the Rothfusz regression equation [67]. Exposure will be examined across gestational windows relevant to fetal development for exploratory analyses. Descriptive statistics will summarize maternal characteristics, environmental exposures, and birth outcomes.

For primary analyses, associations between heat exposure and adverse birth outcomes low birth weight (LBW) and small vulnerable newborns (SVN) will be assessed using multivariable logistic regression for binary outcomes and multivariable linear regression for continuous birth weight. Heat exposure will be modelled primarily as a continuous variable. All models will adjust for maternal age, socioeconomic status, gestational age at delivery, parity, and season. Effect modification by maternal characteristics and season will be examined.

Exploratory analyses will include trimester-specific models to identify sensitive exposure windows. Sensitivity analyses excluding multiple births will assess the robustness of findings among singletons. Alternative exposure definitions will be tested for consistency, including (i) number of days with daily maximum temperature >40°C [68], and (ii) the 90th percentile of the temperature distribution [69]. Exploratory analyses will evaluate additional exposure definitions to determine which metrics demonstrate the strongest associations with outcomes and could be recommended for future use or validation.

Distributed lag and time-varying exposure models will be explored to assess delayed or cumulative effects across gestation. Potential non-linear exposure-response relationships will be examined using Generalized Additive Models (GAMs), with results reported as supplementary to the primary linear models. Given multiple exposure definitions in exploratory analyses, findings will be interpreted cautiously, focusing on effect sizes, confidence intervals, and biological plausibility rather than p-values alone. For a subset of the study participants, mediation analysis will be conducted to investigate potential biological pathways linking heat exposure to fetal growth restriction, focusing on maternal stress response, inflammation, and placental dysfunction. All mediation models will adjust for key confounders. Statistical analyses will be performed using Stata version 18.

Data Quality Assurance

Data will be collected using handheld devices equipped with a dedicated data collection application, enabling real-time capture and secure storage of participant information at enrollment and follow-up. At the end of each day, data will be transmitted via a secure internet connection to the Aga Khan University (AKU) server. In areas where internet access is unavailable, the team leader will export the data manually to a password-protected device to ensure no data is lost. Environmental data from wearable and fixed devices will be retrieved periodically by designated staff and uploaded to the server. All data will be archived in a secure repository with access restricted through AKU LAN authentication, and user access will be managed according to assigned roles. A remote backup system, synchronized daily, will safeguard data against loss or corruption.

To ensure data quality, automated validation checks will be integrated into the data entry platform to flag out-of-range values and inconsistencies, particularly in anthropometric measurements and dietary data. A dedicated sonologist will centrally oversee field-based imaging activities and conduct daily quality assessments of ultrasound, Doppler, and echocardiography data to ensure image clarity and diagnostic accuracy. Standard Operating Procedures (SOPs) will be disseminated to all study teams and strictly followed across all stages, including participant recruitment, data collection, data management, and analysis. Biochemical assays will also adhere to standardized protocols with appropriate internal quality control measures.

Ethical Considerations

The study protocol has been reviewed and approved by the Ethical Review Committee (ERC) of the Aga Khan University and National Bioethics Committee (NBC). Informed consent will be obtained from all participants prior to enrollment. Data confidentiality and participant privacy will be strictly maintained throughout the study.

At each study and follow-up visit, participants will be screened by study physicians for any health issues, including high blood pressure, dehydration, or pregnancy-related complications. Those requiring care will be referred to appropriate healthcare facilities with transportation support. Referral pathways will be in place for managing complications and emergencies at healthcare facilities. Incidental findings, such as cardiac or fetal abnormalities detected during assessments, will be disclosed to participants and referred for specialized care. Pregnancy outcome data will be collected only with participant consent, and all information will be kept confidential.

ELIGIBILITY:
Inclusion Criteria:

* Single or multiple live pregnancy confirmed through ultrasound
* Gestational age less than or equal to 13 weeks and 6 days at enrollment
* At least 18 years of age
* Permanent resident of the study district and plans to deliver within the district
* Willing and able to attend study clinic visits and comply with study procedures throughout pregnancy

Exclusion Criteria:

• Plan to relocate outside the district for more than 3 months during the study period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals who self-identify as women and are currently pregnant are eligible to participate
Study Population: Pregnant women residing in peri-urban and rural areas of the three districts of Sindh, i.e., Matiari, Tharparkar and Tando Muhammad Khan
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Low birthweight (LBW) | Within 48 hours of birth
  Defined as birth weight less than 2,500 grams (5.5 pounds). Newborn weight will be measured within 48 hours of birth using a calibrated Seca 354 infant weighing scale, precise to 0.1 kg. Measurements will be taken independently by two trained anthropometrists. If the difference exceeds 0.05 kg, a third measurement will be taken. Quality assurance procedures and calibration protocols aligned with INTERGROWTH-21st standards will be followed.
  LBW will be analyzed as a binary outcome (Yes/No) to assess its association with prenatal heat stress exposure across different gestational windows.
Incidence of Small Vulnerable Newborns (SVN) births | At the time of delivery
  All live newborns who are either preterm, Small for Gestational Age (SGA), or Low Birth Weight (LBW)

SECONDARY OUTCOMES:
Incidence of Miscarriage | From enrollment till 22 completed weeks of gestation
  Defined as fetal loss before 22 completed weeks of gestation. Gestational age will be confirmed at enrollment using ultrasound measurement of fetal Crown-Rump Length (CRL), with ±7 days accuracy, following INTERGROWTH-21st protocols. It will be assessed as a binary outcome (Yes/No).
Incidence of Pre-term birth | At the time of delivery
  Defined as live birth before 37 completed weeks of gestation. Gestational age will be confirmed at enrollment by study physicians using ultrasound measurement of fetal Crown-Rump Length (CRL), with an accuracy of ±7 days, in accordance with INTERGROWTH-21st standards. Classification will follow standard definitions and will be recorded at the time of delivery. It will be assessed as a binary variable (Yes/No).
Incidence of Small for Gestational Age (SGA) | At the time of delivery
  Description: Defined as neonates born with birth weight below the 10th percentile for gestational age and sex, based on INTERGROWTH-21st standards. Gestational age will be confirmed at enrollment using ultrasound measurement of fetal Crown-Rump Length (CRL), with ±7 days accuracy, following INTERGROWTH-21st protocols. Birth weight will be measured within 48 hours of birth using a Seca 354 infant weighing scale. Classification into term-SGA and preterm-SGA will be based on whether birth occurs before or after 37 completed weeks of gestation. Outcome will be assessed as a binary variable (Yes/No).
Incidence of Stillbirth | From 22 weeks of gestation till birth
  Defined as the birth of a fetus with no signs of life at or after 22 completed weeks of gestation. Data will also be analyzed using a ≥28-week threshold for international comparison. Gestational age will be confirmed by the study physicians through ultrasound using crown rump length (CRL). It will be assessed as a binary outcome (Yes/ No).
Incidence of Gestational Hypertension | From 20 weeks of gestation till birth
  Defined as new-onset systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg, first recorded after 20 weeks of gestation in a previously normotensive woman. It will be measured in mmHg and assessed as a binary variable.
Incidence of Gestational Diabetes Mellitus (GDM) | From enrollment till birth
  Defined as hyperglycemia first detected during pregnancy. Diagnosis will primarily rely on fasting blood glucose >126 mg/dL or random blood glucose >200 mg/dL in the presence of diabetes-related symptoms, measured using point-of-care glucometers by the study physicians at the study clinics. If an oral glucose tolerance test (OGTT) is performed at a registered health facility and shows 2-hour plasma glucose >200 mg/dL, that will also be accepted as diagnostic. All blood glucose measurements will be recorded in mg/dL. GDM will be assessed as a binary outcome (Yes/No).
Incidence of Composite Maternal Morbidity and Mortality (CMMM) | From enrollment till 6 weeks after birth
  Defined as the presence of one or more of the following during pregnancy or within 6 weeks postpartum: 1. postpartum hemorrhage, 2. chorioamnionitis, 3. endometritis, 4. transfusion of ≥2 units of blood, 5. ICU admission, 6. venous thromboembolism, 7. uterine rupture, 8. hysterectomy, 9. cystotomy, 10. ureteral or bowel injury, or 11. maternal death. The outcome will be ascertained and confirmed through clinical diagnosis by the study physicians and health facility records. CMMM will be assessed as a binary outcome (Yes/No).
Composite adverse pregnancy outcomes for the newborn | From enrollment till 7 days after birth
  Includes one or more of the following conditions:
  1. Severe fetal growth restriction (FGR): defined as antenatally diagnosed absent or reversed end-diastolic flow in the umbilical artery; Birth weight < 10th centile and abnormal Doppler ; Birth weight < 3rd centile1 based on INTERGROWTH-21st newborn size standard
  2. Pre-eclampsia with severe features: defined as repeated episodes of severe hypertension despite maintenance treatment with at least two (instead of three as per ISSHP definition) antihypertensive agents, plus pre-eclampsia arising before 34 weeks' gestation according to amended ISSHP criteria
  3. Neonatal death: defined as death < 7 days after birth
  4. Clinical diagnosis of placental abruption
  5. Severe placental lesions: defined as high-grade or severe maternal vascular malperfusion; High-grade/severe fetal vascular malperfusion This composite indicator will be assessed as binary outcome (Yes/No) and each sub-component will also be reported separately.
Incidence of Congenital Fetal Anomalies | From enrollment till birth
  Defined as structural or functional fetal abnormalities identified through obstetric ultrasound scans during pregnancy or postnatally via physical examination or diagnostic imaging. Diagnosis will be confirmed by study physicians. It will be assessed as a Binary outcome (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Jai K Das, MBBS, PhD Public Health, Principal Investigator — Aga Khan University
Locations (3):
- Pakistan (3):
  - Matiari Research and Training Centre, Matiari, Sindh
  - Mithi Study Site Office, Mithi, Sindh
  - Tando Muhammad Khan (TMK) Study Site Office, Tando Muhammad Khan, Sindh

IPD SHARING:
Plan to Share IPD: Undecided